CLINICAL TRIAL: NCT01502852
Title: Identifying the Needs of OEF/OIF Veterans and Their Families: TBI and Co-Occurring Behavioral Health Issues
Brief Title: Identifying the Needs of Operation Enduring Freedom/Operation Iraqi Freedom (OEF/OIF) Veterans and Their Families: TBI and Co-Occurring Behavioral Health Issues
Status: Completed | Type: Observational
Sponsor: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Lisa Brenner, MIRECC Director, VA Eastern Colorado Health Care System
Other Study IDs: 11-0720; PO IHA TBIP1125855 (Other Grant/Funding Number: HRSA)
Record Dates: First submitted 2011-12-29; First posted 2012-01-02 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Traumatic Brain Injury; Co-Occurring Behavioral Health Issues
Keywords: OEF/OIF Veterans; Traumatic Brain Injury; Community Mental Health
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Ecologic or Community
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- OEF/OIF Veterans with TBI
- Family Members and Friends: Family Members and Friends of OEF/OIF Veterans with TBI
- Community Mental Health Center Providers: Community Mental Health Center providers working with OEF/OIF Veterans with TBI

SUMMARY:
The purpose of this study is to explore and potentially increase the capacity of the non-VA community mental health system within the state of Colorado to provide a comprehensive and coordinated service delivery system for Operation Enduring Freedom (OEF)/Operation Iraqi Freedom (OIF) Veterans and their families. The specific population of interest is OEF/OIF Veterans with a history of traumatic brain injury (TBI) and co-occurring behavioral health issues.

DETAILED DESCRIPTION:
The focus of this project is on qualitative data collection to facilitate product development including assessment and treatment guidelines to improve non-VA community mental health care for OEF/OIF Veterans with TBI and co-occurring behavioral health issues within the state of Colorado. In addition to the development of assessment and treatment guidelines, other products developed through this study will include a training and accompanying toolkit, which may be used for annual educational training of mental health providers. As such, there are no hypotheses associated with this study. This statewide initiative may not only improve quality and access to non-VA community mental health care for persons with TBI and co-occurring behavioral health issues within Colorado, but also serve as a model for implementation across the country.

ELIGIBILITY:
Inclusion Criteria:

* Colorado Behavioral Health Organization (BHO) mental health providers
* OEF/OIF United States Veterans
* Family members and/or friends of OEF/OIF United States Veterans
* Ages 18-65

Exclusion Criteria:

- N/A

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: OEF/OIF Veterans with a history of TBI, their family members/friends, and community mental health providers working with these Veterans.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2011-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Focus Groups | One Time

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A Brenner, PhD, Principal Investigator — VISN 19 MIRECC; University of Colorado, School of Medicine, Dept. of Psychiatry
Locations (1):
- VISN 19 MIRECC, Denver VAMC, Denver, Colorado, United States